CLINICAL TRIAL: NCT06077292
Title: Impacts of THC Potency of Cannabis Concentrates and THC Metabolism on Cognitive Impairment in Young Adults
Brief Title: Cannabis THC Potency, Metabolism, and Cognitive Impairment in Young Adults
Acronym: THC-YA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Advocates for Human Potential (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 23-39581
Record Dates: First submitted 2023-10-04; First posted 2023-10-11 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Cannabis Use; THC; Marijuana Use; Cognitive Impairment; THC Vaping
Keywords: Cannabis; Marijuana; High Potency THC; Dabs; Wax; Young Adult; Youth
MeSH Terms: conditions — Marijuana Use; Cognitive Dysfunction; Vaping; Marijuana Abuse

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 15% THC Potency Reduction Group (Experimental): Participants will be incentivized to use THC products that are at least 15% less potent than baseline
  Interventions: Behavioral: 15% THC Potency Reduction
- 35% THC Potency Reduction Group (Experimental): Participants will be incentivized to use THC products that are at least 35% less potent than baseline
  Interventions: Behavioral: 35% THC Potency Reduction

INTERVENTIONS:
Behavioral: 15% THC Potency Reduction — Participants will be incentivized to use THC products that are at least 15% less potent than baseline
  Arms: 15% THC Potency Reduction Group
Behavioral: 35% THC Potency Reduction — Participants will be incentivized to use THC products that are at least 35% less potent than baseline
  Arms: 35% THC Potency Reduction Group

SUMMARY:
The goal of this interventional study is to determine the impact of high potency THC product use on cognitive function of young adults aged 21-25.

The main question it aims to answer is: will cannabis users who switch to less potent THC products demonstrate improved cognitive function compared to baseline?

Other questions this study aims to answer include:

* Can researchers accurately assess THC consumption among frequent cannabis users?
* Can researchers effectively incentivize cannabis users to use less potent THC products?
* Do genetic variations in THC metabolism impact urinary THC excretion?
* Do genetic variations in THC metabolism impact cognitive performance in cannabis users?
* Are quantitative urinary THC values predictive of cognitive impairment?
* How can researchers use research findings to inform harm reduction practices for people who use cannabis?

Participants will submit blood and urine samples and be incentivized to use less potent THC products.

DETAILED DESCRIPTION:
The goal of this interventional study is to determine the impact of high potency THC product use on cognitive function of young adults aged 21-25.

The aims aims of this study are:

1. Evaluate feasibility of assessing THC consumption, genetic variation in THC metabolism, urinary THC excretion, and cognitive performance in users of high potency cannabis products.
2. Test the effectiveness of an incentivization protocol aimed at encouraging cannabis users to use less potent THC products as a means of harm reduction.
3. Compare group differences between the high and low THC-reduction groups on THC metabolism (urine) and cognitive performance while controlling for any changes in frequency and amount of cannabis used.
4. Identify whether participant predisposition to poorly metabolize THC (i.e., CYP2C9*3 carriers vs. others) impacts urinary THC excretion in the experimental condition relative to baseline in both groups.
5. Identify whether participant predisposition to poorly metabolize THC (i.e., CYP2C9*3 carriers vs. others) impacts cognitive performance in the experimental condition relative to baseline in both groups.
6. Determine whether quantitative urinary THC values correlate with measures of cognitive performance.
7. Communicate basic findings regarding relationships between variables and outcomes in the form of a scorecard to help provide harm reduction strategies for youth who use cannabis.

Participants will:

* Undergo a baseline assessment of cognitive performance and will submit blood and urine samples to assess genetic variation in THC metabolism, and baseline urinary THC excretion.
* Be randomized to two groups: 1) lower THC reduction group (incentivized to use THC products that are at least 15% less potent than baseline) and 2) higher THC reduction group (incentivized to use THC products that are at least 35% less potent than baseline) .
* Submit urine samples at baseline and weekly for 5 weeks to measure urinary THC excretion.
* Complete weekly follow up surveys assessing cannabis use patterns, reinforcing value of the cannabis product(s) used, symptoms of cannabis withdrawal, and presence of positive and negative emotions.
* Undergo re-assessment of cognitive performance after 5 weeks of intervention.

Researchers will compare if participants in each group are able to use less potent THC products and whether the use of less potent THC products results in improved cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 21-25
* Resides in San Francisco
* Self-report cannabis concentrate use as their primary method of cannabis use
* Self-report using cannabis daily or almost daily (i.e., at least 6 out of 7 days during each of the last 4 weeks)
* Self-report only purchasing cannabis from regulated retail stores in California.

Exclusion Criteria:

* Pregnant
* Regularly uses other drugs (other than nicotine)

Ages: 21 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2026-03-14 (Estimated); Study Completion 2026-03-14 (Estimated)

PRIMARY OUTCOMES:
Change in Rapid Visual Information Processing Score | Baseline and 5 weeks
  Cognitive performance will be assessed using the CANTAB, a computer-based cognitive assessment system. Participants in this study will complete a battery of seven neuropsychological tests. CANTAB is administered to subjects using a touch screen computer and is language- and culture- independent. Participants scores at 5 weeks will be compared to their baseline scores.
  The Rapid Visual Information Processing test takes 9 minutes to complete and is scored on a scale of 0-54, with a higher score indicative of better cognitive performance.
Change in Paired Associates Learning score | Baseline and 5 weeks
  Cognitive performance will be assessed using the CANTAB, a computer-based cognitive assessment system. Participants in this study will complete a battery of seven neuropsychological tests. CANTAB is administered to subjects using a touch screen computer and is language- and culture- independent. Participants scores at 5 weeks will be compared to their baseline scores.
  The Paired Associates Learning test takes 8 minutes to complete and is scored on a scale of 0-100%, with a higher percentage indicative of better cognitive performance.
Change in Delayed Matching-to-Sample Score | Baseline and 5 weeks
  Cognitive performance will be assessed using the CANTAB, a computer-based cognitive assessment system. Participants in this study will complete a battery of seven neuropsychological tests. CANTAB is administered to subjects using a touch screen computer and is language- and culture- independent. Participants scores at 5 weeks will be compared to their baseline scores.
  The Delayed Matching-to-Sample test takes 7 minutes to complete and is scored on a scale of 0-100%, with a higher percentage indicative of better cognitive performance.
Change in Verbal Recognition Memory score | Baseline and 5 weeks
  Cognitive performance will be assessed using the CANTAB, a computer-based cognitive assessment system. Participants in this study will complete a battery of seven neuropsychological tests. CANTAB is administered to subjects using a touch screen computer and is language- and culture- independent. Participants scores at 5 weeks will be compared to their baseline scores.
  The Verbal Recognition Memory test takes 6 minutes to complete and is scored on a scale of 0-36, with a higher score indicative of better cognitive performance
Change in Spatial Working Memory score | Baseline and 5 weeks
  Cognitive performance will be assessed using the CANTAB, a computer-based cognitive assessment system. Participants in this study will complete a battery of seven neuropsychological tests. CANTAB is administered to subjects using a touch screen computer and is language- and culture- independent. Participants scores at 5 weeks will be compared to their baseline scores.
  The Spatial Working Memory test takes 4 minutes to complete and is scored on a scale of 0-306, with a lower score indicative of fewer errors and better cognitive performance.
Change in One-Touch Stockings of Cambridge score | Baseline and 5 weeks
  Cognitive performance will be assessed using the CANTAB, a computer-based cognitive assessment system. Participants in this study will complete a battery of seven neuropsychological tests. CANTAB is administered to subjects using a touch screen computer and is language- and culture- independent. Participants scores at 5 weeks will be compared to their baseline scores.
  The One-Touch Stockings of Cambridge test takes 10 minutes to complete and scores are based on the time it takes for a participant to solve 20 problems. Shorter time to solve a problem is indicative of better cognitive performance.
Change in Stop Signal Task score | Baseline and 5 weeks
  Cognitive performance will be assessed using the CANTAB, a computer-based cognitive assessment system. Participants in this study will complete a battery of seven neuropsychological tests. CANTAB is administered to subjects using a touch screen computer and is language- and culture- independent. Participants scores at 5 weeks will be compared to their baseline scores.
  The Stop Signal Task test takes 14 minutes to complete and is scored on a scale of 1-1000 milliseconds, with a shorter time indicative of better cognitive performance.

SECONDARY OUTCOMES:
Baseline Urinary THC Excretion | Baseline
  Urinary THC excretion will be measured using liquid chromatography mass spectroscopy (LC/MS/MS). THC levels will be corrected/standardized for level of hydration by dividing total THC by total urine creatinine. Results range from <5 ng/mL to 5,000 ng/mL, with higher values indicative of more THC in the urine.
Week 1 Urinary THC Excretion | 7-10 days after study enrollment.
  Urinary THC excretion will be measured using liquid chromatography mass spectroscopy (LC/MS/MS). THC levels will be corrected/standardized for level of hydration by dividing total THC by total urine creatinine. Results range from <5 ng/mL to 5,000 ng/mL, with higher values indicative of more THC in the urine. Week 1 THC levels will be compared to baseline urine THC levels.
Week 2 Urinary THC Excretion | 14-17 days after study enrollment.
  Urinary THC excretion will be measured using liquid chromatography mass spectroscopy (LC/MS/MS). THC levels will be corrected/standardized for level of hydration by dividing total THC by total urine creatinine. Results range from <5 ng/mL to 5,000 ng/mL, with higher values indicative of more THC in the urine. Week 2 THC levels will be compared to baseline THC levels.
Week 3 Urinary THC Excretion | 21-24 days after study enrollment.
  Urinary THC excretion will be measured using liquid chromatography mass spectroscopy (LC/MS/MS). THC levels will be corrected/standardized for level of hydration by dividing total THC by total urine creatinine. Results range from <5 ng/mL to 5,000 ng/mL, with higher values indicative of more THC in the urine. Week 3 THC levels will be compared to baseline THC levels.
Week 4 Urinary THC Excretion | 28-30 days after study enrollment.
  Urinary THC excretion will be measured using liquid chromatography mass spectroscopy (LC/MS/MS). THC levels will be corrected/standardized for level of hydration by dividing total THC by total urine creatinine. Results range from <5 ng/mL to 5,000 ng/mL, with higher values indicative of more THC in the urine. Week 4 THC levels will be compared to baseline THC levels.
Week 5 Urinary THC Excretion | 35-38 days after study enrollment.
  Urinary THC excretion will be measured using liquid chromatography mass spectroscopy (LC/MS/MS). THC levels will be corrected/standardized for level of hydration by dividing total THC by total urine creatinine. Results range from <5 ng/mL to 5,000 ng/mL, with higher values indicative of more THC in the urine. Week 5 THC levels will be compared to baseline THC levels.

OTHER OUTCOMES:
Urinary THC Excretion in CYP2C9*3 carriers | Baseline
  Predisposition to poorly metabolize THC will be measured at baseline using a blood test to identify carriers of the CYP2C9*3 genetic variant.
  We will then determine whether there are statistically significant differences in baseline and weekly urinary THC levels among CYP2C9*3 carriers compared to non-carriers while controlling for participant reported cannabis use patterns.
Cognitive Performance in CYP2C9*3 carriers | Baseline
  Predisposition to poorly metabolize THC will be measured at baseline using a blood test to identify carriers of the CYP2C9*3 genetic variant.
  We will then determine whether there are statistically significant differences in baseline and 5-week cognitive performance between CYP2C9*3 carriers compared to non-carriers while controlling for participant reported cannabis use patterns.
  Cognitive performance will be assessed using the CANTAB, a computer-based cognitive assessment system. Participants in this study will complete a battery of seven neuropsychological tests. CANTAB is administered to subjects using a touch screen computer and is language- and culture- independent. Participants scores at 5 weeks will be compared to their baseline scores, with lower scores indicating more severe cognitive impairment.
Change in Cannabis Use Disorder Identification Identification Test (CUDIT) score | Baseline and 5 weeks
  Symptoms of a cannabis use disorder will be assessed at baseline using the Cannabis Use Disorder Identification Test (CUDIT). CUDIT scores range from 0 to 32, with a score of 12 or higher indicative of possible cannabis use disorder.
Change in participant reported depression symptoms | Baseline and 5 weeks
  Symptoms of depression will be assessed at baseline and at 5 weeks using the Beck Depression Inventory (BDI). The BDI consists of 21 questions, with scores ranging from 0 to 63; a higher score is indicative of more symptoms of depression. Participant scores at 5 weeks will be compared to their baseline scores.
Baseline Participant Reported Cannabis Use | Baseline
  Participants will complete a baseline survey to determine their pattern of cannabis use one week prior to study enrollment.
  They will be asked to report the brand, name, and THC concentration of the cannabis product(s) they have been using. They will be able to upload photos of product packaging if available.
  They will be asked to report frequency of cannabis use by reporting whether they used their cannabis product in the morning, afternoon, and evening of each of the preceding 7 days.
Week 1 Participant Reported Cannabis Use | 7 days after study enrollment
  Participants will complete a baseline survey to determine their pattern of cannabis use 7 days after study enrollment.
  They will be asked to report the brand, name, and THC concentration of the cannabis product(s) they have been using over the 7 preceding days. They will be asked to upload photos of product packaging.
  They will be asked to report frequency of cannabis use by reporting whether they used their cannabis product in the morning, afternoon, and evening of each of the preceding 7 days.
  THC concentration and frequency of use will be compared to baseline cannabis use.
Week 2 Participant Reported Cannabis Use | 14 days after study enrollment
  Participants will complete a baseline survey to determine their pattern of cannabis use 14 days after study enrollment.
  They will be asked to report the brand, name, and THC concentration of the cannabis product(s) they have been using over the 7 preceding days. They will be asked to upload photos of product packaging.
  They will be asked to report frequency of cannabis use by reporting whether they used their cannabis product in the morning, afternoon, and evening of each of the preceding 7 days.
  THC concentration and frequency of use will be compared to baseline cannabis use.
Week 3 Participant Reported Cannabis Use | 21 days after study enrollment
  Participants will complete a baseline survey to determine their pattern of cannabis use 21 days after study enrollment.
  They will be asked to report the brand, name, and THC concentration of the cannabis product(s) they have been using over the 7 preceding days. They will be asked to upload photos of product packaging.
  They will be asked to report frequency of cannabis use by reporting whether they used their cannabis product in the morning, afternoon, and evening of each of the preceding 7 days.
  THC concentration and frequency of use will be compared to baseline cannabis use.
Week 4 Participant Reported Cannabis Use | 28 days after study enrollment
  Participants will complete a baseline survey to determine their pattern of cannabis use 28 days after study enrollment.
  They will be asked to report the brand, name, and THC concentration of the cannabis product(s) they have been using over the 7 preceding days. They will be asked to upload photos of product packaging.
  They will be asked to report frequency of cannabis use by reporting whether they used their cannabis product in the morning, afternoon, and evening of each of the preceding 7 days.
  THC concentration and frequency of use will be compared to baseline cannabis use.
Week 5 Participant Reported Cannabis Use | 35 days after study enrollment
  Participants will complete a baseline survey to determine their pattern of cannabis use 35 days after study enrollment.
  They will be asked to report the brand, name, and THC concentration of the cannabis product(s) they have been using over the 7 preceding days. They will be asked to upload photos of product packaging.
  They will be asked to report frequency of cannabis use by reporting whether they used their cannabis product in the morning, afternoon, and evening of each of the preceding 7 days.
  THC concentration and frequency of use will be compared to baseline cannabis use.
Baseline Adapted Cannabis Purchase Task | Baseline
  The relative value of cannabis products used by participants during this trial will be assessed using the adaptive cannabis purchase task. Specifically, participants will be asked to report the largest amount of their preferred cannabis product they would "purchase" at a series of price points using visual analog scales. Participants will respond by placing a mark on the line to indicate their purchase amount, and responses will be anchored by 'none' and 'all of it' and will be coded as values 0-100. Higher values are indicative of higher value attributed to the cannabis product being used.
Week 1 Adaptive Cannabis Purchase Task | 7 days after study enrollment
  The relative value of cannabis products used by participants during this trial will be assessed using the adaptive cannabis purchase task. Specifically, participants will be asked to report the largest amount of their preferred cannabis product they would "purchase" at a series of price points using visual analog scales. Participants will respond by placing a mark on the line to indicate their purchase amount, and responses will be anchored by 'none' and 'all of it' and will be coded as values 0-100. Higher values are indicative of higher value attributed to the cannabis product being used.
Week 2 Adaptive Cannabis Purchase Task | 14 days after study enrollment
  The relative value of cannabis products used by participants during this trial will be assessed using the adaptive cannabis purchase task. Specifically, participants will be asked to report the largest amount of their preferred cannabis product they would "purchase" at a series of price points using visual analog scales. Participants will respond by placing a mark on the line to indicate their purchase amount, and responses will be anchored by 'none' and 'all of it' and will be coded as values 0-100. Higher values are indicative of higher value attributed to the cannabis product being used.
Week 3 Adaptive Cannabis Purchase Task | 21 days after study enrollment
  The relative value of cannabis products used by participants during this trial will be assessed using the adaptive cannabis purchase task. Specifically, participants will be asked to report the largest amount of their preferred cannabis product they would "purchase" at a series of price points using visual analog scales. Participants will respond by placing a mark on the line to indicate their purchase amount, and responses will be anchored by 'none' and 'all of it' and will be coded as values 0-100. Higher values are indicative of higher value attributed to the cannabis product being used.
Week 4 Adaptive Cannabis Purchase Task | 28 days after study enrollment
  The relative value of cannabis products used by participants during this trial will be assessed using the adaptive cannabis purchase task. Specifically, participants will be asked to report the largest amount of their preferred cannabis product they would "purchase" at a series of price points using visual analog scales. Participants will respond by placing a mark on the line to indicate their purchase amount, and responses will be anchored by 'none' and 'all of it' and will be coded as values 0-100. Higher values are indicative of higher value attributed to the cannabis product being used.
Week 5 Adaptive Cannabis Purchase Task | 35 days after study enrollment
  The relative value of cannabis products used by participants during this trial will be assessed using the adaptive cannabis purchase task. Specifically, participants will be asked to report the largest amount of their preferred cannabis product they would "purchase" at a series of price points using visual analog scales. Participants will respond by placing a mark on the line to indicate their purchase amount, and responses will be anchored by 'none' and 'all of it' and will be coded as values 0-100. Higher values are indicative of higher value attributed to the cannabis product being used.
Baseline Participant Reported Cannabis Withdrawal Symptoms | Baseline
  Symptoms of cannabis withdrawal will be assessed using the Cannabis Withdrawal Scale (CWS). The CWS consists of 19 questions and assesses withdrawal symptoms as well as the impact of the symptoms on daily activities. The personal experience score ranges from 0-190, with a higher score indicative of more withdrawal symptoms. The negative experience score ranges from 0-190, with a higher number indicative of more negative impact on daily activities.
Week 5 Participant Reported Cannabis Withdrawal Symptoms | 35 days after study enrollment
  Symptoms of cannabis withdrawal will be assessed using the Cannabis Withdrawal Scale (CWS). The CWS consists of 19 questions and assesses withdrawal symptoms as well as the impact of the symptoms on daily activities. The personal experience score ranges from 0-190, with a higher score indicative of more withdrawal symptoms. The negative experience score ranges from 0-190, with a higher number indicative of more negative impact on daily activities.
Baseline Participant Reported Affect | Baseline
  Positive and negative emotions will be assessed using the Positive and Negative Affect Scale (PANAS), which consists of 20 questions, 10 questions assessing positive emotions, and 10 questions assessing negative emotions. Each set of questions is scored on a scale of 10-50, with a higher score indicative of more positive or negative emotions, respectively.
Week 1 Participant Reported Affect | 7 days after study enrollment
  Positive and negative emotions will be assessed using the Positive and Negative Affect Scale (PANAS), which consists of 20 questions, 10 questions assessing positive emotions, and 10 questions assessing negative emotions. Each set of questions is scored on a scale of 10-50, with a higher score indicative of more positive or negative emotions, respectively.
Week 2 Participant Reported Affect | 14 days after study enrollment
  Positive and negative emotions will be assessed using the Positive and Negative Affect Scale (PANAS), which consists of 20 questions, 10 questions assessing positive emotions, and 10 questions assessing negative emotions. Each set of questions is scored on a scale of 10-50, with a higher score indicative of more positive or negative emotions, respectively.
Week 3 Participant Reported Affect | 21 days after study enrollment
  Positive and negative emotions will be assessed using the Positive and Negative Affect Scale (PANAS), which consists of 20 questions, 10 questions assessing positive emotions, and 10 questions assessing negative emotions. Each set of questions is scored on a scale of 10-50, with a higher score indicative of more positive or negative emotions, respectively.
Week 4 Participant Reported Affect | 28 days after study enrollment
  Positive and negative emotions will be assessed using the Positive and Negative Affect Scale (PANAS), which consists of 20 questions, 10 questions assessing positive emotions, and 10 questions assessing negative emotions. Each set of questions is scored on a scale of 10-50, with a higher score indicative of more positive or negative emotions, respectively.
Week 5 Participant Reported Affect | 35 days after study enrollment
  Positive and negative emotions will be assessed using the Positive and Negative Affect Scale (PANAS), which consists of 20 questions, 10 questions assessing positive emotions, and 10 questions assessing negative emotions. Each set of questions is scored on a scale of 10-50, with a higher score indicative of more positive or negative emotions, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Veronika Mesheriakova, MD, Principal Investigator — University of California, San Francisco; Michael Sofis, PhD, Principal Investigator — Cannabis Public Policy Consulting
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sachse-Seeboth C, Pfeil J, Sehrt D, Meineke I, Tzvetkov M, Bruns E, Poser W, Vormfelde SV, Brockmoller J. Interindividual variation in the pharmacokinetics of Delta9-tetrahydrocannabinol as related to genetic polymorphisms in CYP2C9. Clin Pharmacol Ther. 2009 Mar;85(3):273-6. doi: 10.1038/clpt.2008.213. Epub 2008 Nov 12. PMID 19005461
- [Background] Murray RM, Quigley H, Quattrone D, Englund A, Di Forti M. Traditional marijuana, high-potency cannabis and synthetic cannabinoids: increasing risk for psychosis. World Psychiatry. 2016 Oct;15(3):195-204. doi: 10.1002/wps.20341. PMID 27717258
- [Background] Ramaekers JG, Kauert G, van Ruitenbeek P, Theunissen EL, Schneider E, Moeller MR. High-potency marijuana impairs executive function and inhibitory motor control. Neuropsychopharmacology. 2006 Oct;31(10):2296-303. doi: 10.1038/sj.npp.1301068. Epub 2006 Mar 29. PMID 16572123
- [Background] D'Souza DC, Ganesh S, Cortes-Briones J, Campbell MH, Emmanuel MK. Characterizing psychosis-relevant phenomena and cognitive function in a unique population with isolated, chronic and very heavy cannabis exposure. Psychol Med. 2020 Oct;50(14):2452-2459. doi: 10.1017/S0033291719002721. Epub 2019 Oct 16. PMID 31615592
- [Background] Bidwell LC, Martin-Willett R, Karoly HC. Advancing the science on cannabis concentrates and behavioural health. Drug Alcohol Rev. 2021 Sep;40(6):900-913. doi: 10.1111/dar.13281. Epub 2021 Mar 30. PMID 33783029
- [Background] Bourque J, Potvin S. Cannabis and Cognitive Functioning: From Acute to Residual Effects, From Randomized Controlled Trials to Prospective Designs. Front Psychiatry. 2021 Jun 10;12:596601. doi: 10.3389/fpsyt.2021.596601. eCollection 2021. PMID 34177633